CLINICAL TRIAL: NCT04216147
Title: Percutaneous Needle Electrolysis Versus Surgery in the Treatment of Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, Jose Antonio Garcia Vidal, Doctor, Universidad de Murcia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01/2014
Record Dates: First submitted 2019-12-28; First posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Carpal Tunnel Syndrome
Keywords: carpal tunnel syndrome; nerve compression syndrome; median nerve; physical therapy technique; percutaneous needle electrolysis
MeSH Terms: conditions — Carpal Tunnel Syndrome; Nerve Compression Syndromes | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PNE group (Experimental): Patients received 4 sessions, separated one week between them. The treatment consisted the application of a galvanic current through an acupuncture needle (0,30x30mm). The approach were performed with a transverse axis with a needle in plane, being superficial and deep interface of medium nerve the target tissue. The parameters will be 2 mA (milliamps), 10 seconds, 3 impacts (3: 3: 3).
  Interventions: Other: PNE
- Surgery group (Experimental): Patients received surgery for median nerve release.
  Interventions: Procedure: Surgery for CTS

INTERVENTIONS:
Other: PNE — Percutaneous Needle Electrolysis: the application of galvanic current through an acupuncture needle.
  Arms: PNE group
Procedure: Surgery for CTS — Median nerve release
  Arms: Surgery group

SUMMARY:
The aim of this study is to compare the effectiveness of Percutaneous Needle Electrolysis (PNE) versus surgical treatment in the treatment of Carpal Tunnel Syndrome (CTS).

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years.
* CTS diagnosed by Electromyography (EMG)
* Symptoms of CTS + EMG

Exclusion Criteria:

* Difficulty expressing your feelings properly
* Unsurpassed fear of needles
* History of adverse reactions to needles
* Epilepsy and / or allergies to metals.
* Difficulty expressing your feelings properly
* Existence of diffuse peripheral neuropathy or cervical radiculopathy
* History of potential concurrent cause of idiopathic CTS (such as diabetes, thyroid, chronic rheumatoid arthritis, renal failure with hemodialysis, pregnancy..)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Changes of the Boston Questionnaire for Carpal Tunnel Syndrome | Baseline and after treatments: 6 weeks, 3 months, 6 months and 12 months
  11-question patient-administered survey that rates the severity of the patient's carpal tunnel syndrome-specific symptoms on a scale of 1 (no symptoms) to 5 (worst symptoms)

SECONDARY OUTCOMES:
Changes of the Clinical Symptoms Carpal Tunnel Syndrome Scale | Baseline and after treatments: 6 weeks, 3 months, 6 months and 12 months
  Describe the symptoms of the hand and wrist (pointing to them in a drawing), and using scales of 1 to 5 (1= No difficulty to do it; 5= I can´t do it), measure the difficulty of performing certain activities (writing, buttoning, holding a book ...)
Change of pain level | Baseline and after treatments: 6 weeks, 3 months, 6 months and 12 months
  Visual Analogue Scale (VAS: 0=no pain; 100= pain as bad as can be)
Change of Semmes Weinstein Mini monofilament kit | Baseline and after treatments: 6 weeks, 3 months, 6 months and 12 months
  Contact threshold, to assess if there is a decrease in sensitivity
Change of the Hand Dynamometer | Baseline and after treatments: 6 weeks, 3 months, 6 months and 12 months
  Hand grip force
Changes of the Muscles strength by Kendall´s scale | Baseline and after treatments: 6 weeks, 3 months, 6 months and 12 months
  Muscular strength of Opponens pollicis and Abductors policies. Scale of 0 to 5 (0=No visible or palpable contraction; 5=Full ROM against gravity, maximum resistance)
Changes of the SF-12 Questionnaire (Short Form 12 Questionnaire) | Baseline and after treatments: 6 weeks, 3 months, 6 months and 12 months
  12 questions self-administered. Assess quality of life, general health and well-being using scales of 1 to 5 (1= Ever; 5= Never)

OTHER OUTCOMES:
Direct and indirect health cost measures | 12 months after treatments
  Number of visits to the specialist, number of hospitalization days, number of physiotherapy sessions, prescribed medication, days of work absenteeism

IPD SHARING:
Plan to Share IPD: No